CLINICAL TRIAL: NCT06234215
Title: Functional Task Training Combined With Electrical Stimulation on Balance and Motor Abilities in Children With Diplegia
Brief Title: Effect of Electrical Stimulation With Functional Task Training on Balance and Motor Abilities in Children With Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Randa Adel, specialist physiotherapy Randa Adel Mousa Mostafa Mousa, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E.S and balance in diplegia
Record Dates: First submitted 2024-01-05; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group had functional task training (Active Comparator): this group doing functional task training exercise for 50 min 3 times per week for two months
  Interventions: Other: functional task training
- study group had functional task training combined with electrical stimulation (Experimental): this group doing functional task training exercise combined with electrical stimulation for 50 min 3 times per week for two months
  Interventions: Device: functional electrical stimulation; Other: functional task training

INTERVENTIONS:
Device: functional electrical stimulation — electrical stimulation during function
  Arms: study group had functional task training combined with electrical stimulation
Other: functional task training — functional exercise

SUMMARY:
The aims of the study are to:

1. Investigate the combined effect of functional task training with electrical stimulation of bilateral hip abductor muscles on balance in children with diplegia.
2. Investigate the combined effect of functional task training with electrical stimulation of bilateral hip abductor muscles on motor abilities in children with diplegia.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of permanent disorders of movement and posture. It is non-progressive lesion or abnormality of immature brain. The term cerebral refers to the brain and palsy refers to the loss or impairment of motor function.

Functional electrical stimulation (FES) is a subtype of neuromuscular electrical stimulation (NMES) in which the stimulation assists functional and purposeful movements. This is achieved by applying electrical stimulation to muscles that, when they contract, produce a movement that can be used functionally.The FES is used to provide electrical stimulation via the peripheral nervous system to activate muscle contractions to assist functional activities when nervous or musculo-skeletal systems are damaged.The common applications of FES include strengthening muscle, reducing muscle spasticity, increasing range of motion, improving upper extremity function and walking speed.

ELIGIBILITY:
Inclusion Criteria:

* Their ages will range from 7-11 years.
* Both genders will be included.
* Their degree of spasticity will range from 1 to 1+ according to Modified Ashworth Scale (Meseguer-Henarejos et al., 2018).
* Their motor function will be at level I & II according to Gross Motor Function --- -Classification system (Palisano et al., 2008).
* They will be understanding instructions.

Exclusion Criteria:

* Children will be excluded from the study if they have any of the following criteria:

Musculoskeletal fixed deformities in upper limb, lower limb or spine.

* Visual or hearing problems.
* Epilepsy.
* Botulinium toxin therapy or orthopedic surgery within the past 6months or within the study period.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Humac balance system | two months
  static and dynamic balance when values inscrease the results are better.

SECONDARY OUTCOMES:
Growth motor functional scale | two months
  measuring motor abilities standing and walking when values increase the results are better.

CONTACTS AND LOCATIONS:
Overall Officials: ‪Randa Adel‬, master, Principal Investigator — Cairo University
Locations (1):
- ‪Randa Adel‬, Ītāy al Bārūd, El-beheira, Egypt